CLINICAL TRIAL: NCT00003092
Title: Clinical Pharmacology of Paclitaxel in Relation to Patient Age
Brief Title: Paclitaxel in Treating Older Patients With Solid Tumors
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-9762; U10CA031946 (NIH); CLB-9762; CDR0000065800 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-07

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Paclitaxel (Experimental): Patients receive a single dose of IV paclitaxel over 3 hours. Additional cycles of paclitaxel will be given at the discretion of the physician.
  Patients are followed for second malignancies, disease progression, and survival.
  Interventions: Drug: paclitaxel

INTERVENTIONS:
Drug: paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase III trial to study the effectiveness of paclitaxel in treating older patients who have solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine whether there is a relationship between pharmacokinetic measurements of paclitaxel and aging.
* Determine whether there is a relationship between the toxic effects of paclitaxel and aging.

OUTLINE: Patients are stratified according to age (cohort 1: patients 55 to 64 vs cohort 2: patients 65 to 75 vs cohort 3: patients 75 and over).

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven nonhematologic malignancy

PATIENT CHARACTERISTICS:

Age:

* 55 and over

Performance status:

* Zubrod 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Granulocyte count at least 1,500/mm3
* Platelet count at least 100,000/mm3

Hepatic:

* Bilirubin less than 1.5 mg/dL
* SGOT less than 2.0 times upper limit of normal (ULN)

Renal:

* Creatinine no greater than 1.5 times ULN

Cardiovascular:

* No uncontrolled or severe cardiovascular disease

Other:

* No serious intercurrent medical illnesses that in the judgement of the investigator compromise patient care
* No psychiatric conditions that would preclude study
* No requirement for antibiotics for active acute infection

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin)
* No more than one prior chemotherapy regimen allowed
* No prior paclitaxel allowed

Endocrine therapy:

* Not specified

Radiotherapy:

* At least 4 weeks since prior radiation therapy

Surgery:

* Not specified

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 1997-09; Primary Completion 2006-03 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Overall survival | Up to 5 years
Disease-free progression | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Stuart M. Lichtman, MD, Study Chair — Don Monti Comprehensive Cancer Center at North Shore University Hospital
Locations (32):
- United States (32):
  - Rebecca and John Moores UCSD Cancer Center, La Jolla, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - CCOP - Christiana Care Health Services, Wilmington, Delaware
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Marlene and Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center - University Campus, Worcester, Massachusetts
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Ellis Fischel Cancer Center - Columbia, Columbia, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - Roswell Park Cancer Institute, Buffalo, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - North Shore University Hospital, Manhasset, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - New York Presbyterian Hospital - Cornell Campus, New York, New York
  - Mount Sinai Medical Center, NY, New York, New York
  - State University of New York - Upstate Medical University, Syracuse, New York
  - CCOP - Syracuse Hematology-Oncology Associates of Central New York, P.C., Syracuse, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Rhode Island Hospital, Providence, Rhode Island
  - University of Tennessee Cancer Institute, Memphis, Tennessee
  - Vermont Cancer Center, Burlington, Vermont
  - MBCCOP - Massey Cancer Center, Richmond, Virginia

REFERENCES:
- [Result] Lichtman SM, Hollis D, Miller AA, Rosner GL, Rhoades CA, Lester EP, Millard F, Byrd J, Cullinan SA, Rosen DM, Parise RA, Ratain MJ, Egorin MJ; Cancer and Leukemia Group B (CALGB 9762). Prospective evaluation of the relationship of patient age and paclitaxel clinical pharmacology: Cancer and Leukemia Group B (CALGB 9762). J Clin Oncol. 2006 Apr 20;24(12):1846-51. doi: 10.1200/JCO.2005.03.9289. Epub 2006 Mar 27. PMID 16567769
- [Result] Lichtman SM, Egorin M, Rosner G, et al.: Clinical pharmacology of paclitaxel in relation to patient age: CALGB 9762. [Abstract] Proceedings of the American Society of Clinical Oncology 18: A732, 1999.